CLINICAL TRIAL: NCT05968040
Title: Point Of Care Ultrasound For Prediction Of Fluid Responsiveness in Off Pump Coronary Artery Bypass Grafting Surgery, Comparison Between Carotid Doppler Peak Velocity And IVC Distensibility Index
Brief Title: Point Of Care Ultrasound For Prediction Of Fluid Responsiveness in Off Pump Coronary Artery Bypass Grafting Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ain shams H.
Record Dates: First submitted 2023-07-16; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Prevention of Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- responder (Active Comparator)
  Interventions: Procedure: Inferior vena cava diameter measurement by ultrasonography; Procedure: difference between peak velocities of carotid artery by ultrasound; Procedure: cardiac output be transthoracic echocardiography
- non responder (Active Comparator)
  Interventions: Procedure: Inferior vena cava diameter measurement by ultrasonography; Procedure: difference between peak velocities of carotid artery by ultrasound; Procedure: cardiac output be transthoracic echocardiography

INTERVENTIONS:
Procedure: Inferior vena cava diameter measurement by ultrasonography — The diameter of the inferior vena cava will be measured at 2 cm close to the entrance of the right atrium. Ultrasound images will be taken at the end of inspiration (Dmax) and at the end expiration (Dmin) to calculate the inferior vena cava dispensability index (dIVC), and will be recorded before and after fluid challenge test of 5 ml/kg crystalloid within 15 min. The IVC distensibility index (IVC-DI) will be calculated using the formula: IVC-DI = IVCmax - IVCmin/ IVCmin. The indices will be expressed as a percentage.
Procedure: difference between peak velocities of carotid artery by ultrasound — Carotid ultrasound images will be obtained from the left CCA in both short-axis and long-axis views by experienced sonographers. The patient will be in supine position, with the head rotated slightly to the right. A broadband linear array transducer 12-4 MHz and the short-axis view will be used for orientation and identification of the CCA. Next, in the long-axis view, Peak Waveform Doppler signals will be acquired by placing a 0.5 mm calliper at the center of the vessel and parallel to the vessel walls, approximately 2 cm proximal from the carotid bifurcation. Insonation-angles between the ultrasound beam and blood flow will be maintained.
  ΔVpeakCCA = (MaxCDPV-MinCDPV)+(MaxCDPV+MinCDPV)x100
Procedure: cardiac output be transthoracic echocardiography — CO will be recorded as baseline measure and after fluid administration. If CO increased more than 15%, it will be considered fluid responder. Increase in cardiac output = (cardiac output after first fluid challenge - cardiac output before)/cardiac output before) X 100.
  TTE will be used to measure LTOT and VTI x HR.

SUMMARY:
To exclude hypovolemia before starting off pump coronary artery grafting surgeries by an efficient and good predictive test. We will assess the sensitivity and specificity of dynamic IVC-derived parameters (dispensability index) in comparison to carotid Doppler peak velocity as predictors of fluid response before skin incision in patients undergoing off Pump cardiac surgery.

DETAILED DESCRIPTION:
Monitoring We will monitor all patients using, invasive blood pressure, pulse oximeter, central venous pressure (CVP), 5 leads Electrocardiogram ECG and capnogram.

Anesthetic technique:

Anesthesia will be inducted by; lidocaine 1.5 mg/Kg, fentanyl 10 mic/kg, propofol (2 mg/kg) and atracurium (0.5 mg/kg). After good muscle relaxation, intubation will be done smoothly. Mechanical ventilation parameters will be fixed in all patients during the study period. Tidal volume will be adjusted to 10 ml/kg without positive end expiration pressure. End tidal carbon dioxide will be kept around 35-40 centimeter water(cmH2O). Anesthesia will be maintained by Sevoflurane 2% minimal alveolar concentration(MAC), atracurium infusion; 0.05-0.01 mg/kg/min and fentanyl infusion rate; 1 mic/kg/hour.

Study measurements:

After induction of anesthesia we will perform the measurement of the diameter of the inferior vena cava through standard ultrasonic techniques. The M-mode portable ultrasound 1-5 megahertz (MHz) transthoracic phased-array transducer probe will be positioned longitudinally along the xiphoid process when the patient is supine. The diameter of the inferior vena cava will be measured at 2 cm close to the entrance of the right atrium. Ultrasound images will be taken at the end of inspiration (Dmax) and at the end expiration (Dmin) to calculate the inferior vena cava dispensability index (dIVC), and will be recorded before and after fluid challenge test of 5 ml/kg crystalloid within 15 min. The inferior vena cava (IVC) distensibility index (IVC-DI) will be calculated using the formula: IVC-DI = IVCmax - IVCmin/ IVCmin. The indices will be expressed as a percentage.

Carotid ultrasound images will be obtained from the left common carotid artery( CCA) in both short-axis and long-axis views by experienced sonographers. The patient will be in supine position, with the head rotated slightly to the right. A broadband linear array transducer 12-4 MHz and the short-axis view will be used for orientation and identification of the CCA. Next, in the long-axis view, Peak Waveform Doppler signals will be acquired by placing a 0.5 mm calliper at the center of the vessel and parallel to the vessel walls, approximately 2 cm proximal from the carotid bifurcation. Insonation-angles between the ultrasound beam and blood flow will be maintained.

difference of peak velocity(ΔVpeak) of CCA = (MaxCDPV-MinCDPV)+(MaxCDPV+MinCDPV)x100 2

cardiac output (CO) will be recorded as baseline measure and after fluid administration. If CO increased more than 15%, it will be considered fluid responder. Increase in cardiac output = (cardiac output after first fluid challenge - cardiac output before)/cardiac output before) X 100.

Transthoracic echocardiography(TTE) will be used to measure LTOT and velocity time integral (VTI) x heart rate (HR).

CVP, mean arterial pressure, pulse pressure, difference between diameters of IVC during inspiration and expiration (ΔIVC-d) in single respiratory cycle, and difference between velocities of carotid Doppler peak velocity in single respiratory cycle (ΔCDPV) will all be measured as hemodynamic records.

The benefits include declining heart rate, normotension, and increase and urine volume, also known as fluid responsiveness

ELIGIBILITY:
Inclusion Criteria:

* Patients with accepted cardiac capacity (EF >45%)
* Patients scheduled for off pump open heart surgeries for coronary artery grafting

Exclusion Criteria:

* age under 18 years,
* patients with poor cardiac capacity
* patients suffering any type of arrhythmias
* preoperative left ventricular dilatation (end-diastolic dimension ≥6 cm)
* preoperative severe tricuspid valve regurgitation,
* preoperative right ventricular dysfunction
* patients with high intrathoracic pressure e.g.chronic obstructive pulmonary disease (COPD).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
cardiac output by transthoracic echocardiography | immediately before fluid administration
  cardiac output = stroke volume x heart rate
cardiac outputby transthoracic echocardiography | immediately after fluid administration
  cardiac output = stroke volume x heart rate

SECONDARY OUTCOMES:
inferior vena cava diameter by ultrasonography | immediately before fluid administration
inferior vena cava diameter by ultrasonography | immediately after fluid administration
carotid peak velocity by ultrasound | immediately before fluid administration
carotid peak velocity by ultrasound | immediately after fluid administration
central venous pressure measurement | immediately before fluid administration
central venous pressure measurement | immediately after fluid administration
mean blood pressure | immediately before fluid administration
mean blood pressure | immediately after fluid administration
heart rate | immediately before fluid administration
heart rate | immediately after fluid administration
usage of ionotropic support (adrenalin, noreadrenalin,dopamine and dubotamine) | during the intraoperative period

IPD SHARING:
Plan to Share IPD: No